CLINICAL TRIAL: NCT01226732
Title: A Phase I Study of the Hsp90 Inhibitor AUY922 Plus Capecitabine for the Treatment of Patients With Advanced Solid Tumors
Brief Title: A Study of the Hsp90 Inhibitor AUY922 Plus Capecitabine for the Treatment of Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 143
Record Dates: First submitted 2010-10-18; First posted 2010-10-22 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Metastatic or Unresectable Solid Tumor Malignancy
Keywords: Solid tumor; Capecitabine; Hsp90 inhibitor AUY922
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Dose Level 1 (Experimental): Hsp90 Inhibitor AUY922: 22mg/m2 IV days 1, 8, and 15 of 21-day cycles Capecitabine: 1000mg/m2 PO BID d 1-14 of 21-day cycles
  Interventions: Drug: Capecitabine; Drug: Hsp90 Inhibitor AUY 922
- Dose Level 2 (Experimental): Hsp90 Inhibitor AUY922: 28mg/m2 IV days 1, 8, and 15 of 21-day cycles Capecitabine: 1000mg/m2 PO BID d 1-14 of 21-day cycles
  Interventions: Drug: Capecitabine; Drug: Hsp90 Inhibitor AUY 922
- Dose Level 3 (Experimental): Hsp90 Inhibitor AUY922: 40mg/m2 IV days 1, 8, and 15 of 21-day cycles Capecitabine: 1000mg/m2 PO BID d 1-14 of 21-day cycles
  Interventions: Drug: Capecitabine; Drug: Hsp90 Inhibitor AUY 922
- Dose Level 4 (Experimental): Hsp90 Inhibitor AUY922: 55mg/m2 IV days 1, 8, and 15 of 21-day cycles Capecitabine: 1000mg/m2 PO BID d 1-14 of 21-day cycles
  Interventions: Drug: Capecitabine; Drug: Hsp90 Inhibitor AUY 922
- Dose Level 5 (Experimental): Hsp90 Inhibitor AUY922: 70mg/m2 IV days 1, 8, and 15 of 21-day cycles Capecitabine: 1000mg/m2 PO BID d 1-14 of 21-day cycles
  Interventions: Drug: Capecitabine; Drug: Hsp90 Inhibitor AUY 922
- Dose Level 6 (Experimental): Hsp90 Inhibitor AUY922: 70mg/m2 IV days 1, 8, and 15 of 21-day cycles Capecitabine: 1250mg/m2 PO BID d 1-14 of 21-day cycles
  Interventions: Drug: Capecitabine; Drug: Hsp90 Inhibitor AUY 922

INTERVENTIONS:
Drug: Capecitabine — Taken orally twice daily on Days 1 through 14 of 21 day cycle.
  Other Names: Xeloda
Drug: Hsp90 Inhibitor AUY 922 — IV infusion over 60 minutes on Days 1, 8, and 15 of each 21 day cycle

SUMMARY:
The investigators propose this Phase I trial of the combination of AUY922 and capecitabine to determine the maximum tolerated dose (MTD) in patients with advanced solid tumors. This combination treatment has potential applicability in tumor types where capecitabine or fluorouracil is a treatment option, including colorectal and breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic or unresectable solid tumor malignancy that is incurable and for which capecitabine is clinically appropriate.
2. Patient must be ≥4 weeks from administration of last dose of cancer therapy (including radiation therapy, biologic therapy, hormonal therapy or chemotherapy). Patients who received a small molecule targeted therapy as part of their first line treatment regimen must be ≥4 weeks or ≥5 half lives from administration of last dose whichever is shorter. The patient must have recovered from or come to a new chronic stable baseline from all treatment-related toxicities.
3. Eastern Collaborative Oncology Group (ECOG) performance status 0 to 1 (see Appendix A).
4. Life expectancy of ≥3 months.
5. At least one unidimensional measurable lesion definable by MRI or CT scan. Disease must be measurable per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria (see Section 9).
6. Normal bone marrow function defined as:

   * Absolute neutrophil count (ANC) ≥1500/μL
   * Hemoglobin (Hgb) ≥9 g/dL
   * Platelets ≥100,000/μL
7. Adequate hepatic function defined as:

   * AST or ALT and alkaline phosphatase (ALP) must be ≤3 x ULN, or ≤5 x ULN in patients with liver metastases
   * Total bilirubin ≤1.5 x the institutional ULN
8. Renal function defined as:

   • Serum creatinine ≤1.5 x ULN or 24-hour creatinine clearance ≥40 mL/min
9. Normal electrolytes defined as:

   * Phosphorous ≥ LLN
   * Magnesium ≥ LLN
10. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test performed within 7 days prior to start of treatment. Women of childbearing potential must use effective birth control measures during treatment and during the 6 months following completion of study treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately.
11. Must be ≥18 years of age.
12. Patients must be accessible for treatment and follow-up.
13. Patients must be able to understand the investigational nature of this study and give written informed consent prior to study entry.

Exclusion Criteria:

1. Untreated CNS metastases. Patients with treated CNS metastases may be enrolled, provided the patient is asymptomatic, and the patient does not require antiepileptic drugs or steroids as treatment for the CNS metastases.
2. Treatment with therapeutic doses of coumarin-type anticoagulants (maximum daily dose of 1 mg allowed for port line patency permitted).
3. Impaired cardiac function with any one of the following:

   * History (or family history) of long QT syndrome
   * Mean QTc ≥450 msec on baseline ECG
   * History of clinically manifested ischemic heart disease (i.e. myocardial infarction and/or unstable angina) ≤6 months prior to study start
   * History of heart failure or left ventricular (LV) dysfunction (LVEF ≤45%) by MUGA or ECHO
   * Clinically significant ECG abnormalities including 1 or more of the following: left bundle branch block (LBBB), right bundle branch block (RBBB) with left anterior hemiblock (LAHB). ST segment elevation or depression > 1mm, or 2nd (Mobitz II), or 3rd degree AV block.
   * History or presence of atrial fibrillation, atrial flutter or ventricular arrhythmias including ventricular tachycardia or Torsades de Pointes
   * Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
   * Clinically significant resting bradycardia (< 50 beats per minute)
   * Patients who are currently receiving treatment with any medication which has a relative risk of prolonging the QTcF interval or inducing Torsades de Pointes and cannot be switched to an alternative drug or discontinued prior to commencing AUY922 (see Appendix D).
   * Obligate use of a cardiac pacemaker
4. Impairment of gastrointestinal function or gastrointestinal disease that in the opinion of the Investigator may significantly alter the absorption of study drugs (e.g., Crohn's disease, ulcerative disease, uncontrolled vomiting, diarrhea, or malabsorption syndrome).
5. Patients with known diagnosis of human immunodeficiency virus (HIV), hepatitis C virus, or acute or chronic hepatitis B infection.
6. Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Women who are pregnant (positive pregnancy test) or lactating.
8. Any condition that would prevent patient comprehension of the nature of, and risk associated with, the study, and the inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-11; Primary Completion 2013-07 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna C Bendell, MD, Study Chair — SCRI Development Innovations, LLC
Locations (3):
- United States (3):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Oklahoma University, Oklahoma City, Oklahoma
  - Tennessee Oncology, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6
Started | 3 | 3 | 3 | 5 | 3 | 6
Completed | 0 (Patients remained on-study until disease progression or intolerable toxicity) | 0 (Patients remained on-study until disease progression or intolerable toxicity) | 0 (Patients remained on-study until disease progression or intolerable toxicity) | 0 (Patients remained on-study until disease progression or intolerable toxicity) | 0 (Patients remained on-study until disease progression or intolerable toxicity) | 0 (Patients remained on-study until disease progression or intolerable toxicity)
Not Completed | 3 | 3 | 3 | 5 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 6 | 23
Age, Continuous [Median (Full Range); unit: years] | 59 [53 to 66] | 51 [37 to 64] | 64 [45 to 65] | 60 [47 to 68] | 58 [49 to 63] | 65.5 [54 to 71] | 60 [37 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 2 | 1 | 3 | 7
  Male | 3 | 3 | 2 | 3 | 2 | 3 | 16
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 5 | 3 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: Dose Determination
Description: To determine the maximum tolerated dose (MTD) of AUY922 plus capecitabine in patients with advanced solid tumors.
Time Frame: 18 months
Measure: Number; unit: mg/m^2
Groups:
- All Patients: The Maximum Tolerated Dose (MTD) is determined for all patients
Arm/Group | All Patients
Number analyzed (Participants) | 23
mg/m^2
  AUY922 dose | 70
  Capecitabine dose | 1250

2. Secondary Outcome: Drug Related Toxicities
Description: To evaluate the drug related toxicities associated with different doses of the drugs used in this regimen.
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 6
participants
  Vision changes | 0 | 0 | 1 | 3 | 3 | 6
  Diarrhea | 1 | 1 | 2 | 3 | 3 | 4
  Fatigue | 3 | 0 | 1 | 1 | 1 | 4
  Nausea | 2 | 2 | 1 | 3 | 1 | 0
  Hand-foot syndrome | 1 | 0 | 0 | 2 | 1 | 5
  Anorexia | 2 | 0 | 0 | 3 | 1 | 2
  Vomiting | 2 | 0 | 1 | 2 | 2 | 0

3. Secondary Outcome: Preliminary Efficacy Assessment: Response Rate (RR)
Description: Response Rate (RR) is defined as the total number of patients with Complete Response (CR) or Partial Response (PR) as defined in RECIST v2. CR is defined as the dissappearance of all target lesions, disappearance of all non-target lesions and normalization of tumor markers. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: 18 months
Population: Includes all patients evaluable for response. 4 patients were not evaluable: dose level 2 (1 pt), dose level 4 (2 pts), dose level 6 (1 pt).
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 5
participants | 1 | 0 | 0 | 2 | 1 | 0

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/3 | 1/5 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 5/5 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=3) | Dose Level 4 (N=5) | Dose Level 5 (N=3) | Dose Level 6 (N=6)
General disorders and administration site conditions - Other, failure to thrive (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=3) | Dose Level 4 (N=5) | Dose Level 5 (N=3) | Dose Level 6 (N=6)
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 2 | 4 | 2 | 5
Nausea (Gastrointestinal disorders) | 2 | 2 | 1 | 5 | 2 | 2
Fatigue (General disorders) | 3 | 0 | 1 | 3 | 1 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 4 | 1 | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 1 | 5
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 1 | 2
Eye disorders - Other, vision changes (Eye disorders) | 0 | 0 | 1 | 1 | 2 | 2
Mucositis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 0 | 0
Edema limbs (General disorders) | 2 | 0 | 0 | 1 | 0 | 1
Floaters (Eye disorders) | 0 | 0 | 0 | 1 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 1
Weight loss (Investigations) | 1 | 0 | 0 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 2
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Flashing lights (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 2
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1
Skin and subcutaneous tissue disorders - Other, skin changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blurred vision (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Eye disorders - Other, color differentiation difficulties (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites